CLINICAL TRIAL: NCT06952907
Title: Femoral Versus Radial Artery Catheterization for Invasive Arterial Pressure Monitoring in Cardiac Surgery Patients: the FERARI Randomized Superiority Study
Brief Title: Femoral Versus Radial Invasive Arterial Pressure Monitoring in Cardiac Surgery Patients
Acronym: FERARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guillaume BESCH (Other)
Responsible Party: Sponsor-Investigator, Guillaume BESCH, Professor of Anesthesiology and Intensive Care Medicine, Centre Hospitalier Universitaire de Besancon
Organization: Centre Hospitalier Universitaire de Besancon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/897
Record Dates: First submitted 2025-04-18; First posted 2025-05-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Vasoplegia Syndrome; Vasoplegia; Cardiac Surgical Procedures; Arterial Pressure; Hypotension During Surgery; Hypotension Postprocedural; Norepinephrine
Keywords: Invasive arterial blood pressure monitoring; Vasoplegia syndrome; Cardiac surgery; Norepinephrine
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral group (Active Comparator): Patients in the femoral group undergo femoral artery catheterization for continuous invasive arterial blood pressure monitoring.
  Interventions: Other: Femoral artery catheterization for continuous invasive arterial blood pressure monitoring
- Radial group (Active Comparator): Patients in the arterial group undergo arterial artery catheterization for continuous invasive arterial blood pressure monitoring.
  Interventions: Other: Radial artery catheterization for continuous invasive arterial blood pressure monitoring

INTERVENTIONS:
Other: Femoral artery catheterization for continuous invasive arterial blood pressure monitoring — Femoral artery catheterization allow for continuous invasive arterial blood pressure monitoring.
  Arms: Femoral group
Other: Radial artery catheterization for continuous invasive arterial blood pressure monitoring — Radial artery catheterization allows for continuous invasive arterial blood pressure monitoring
  Arms: Radial group

SUMMARY:
Background: Acute circulatory failure, often presenting as arterial hypotension, is a major contributor to postoperative morbidity and mortality. Accurate blood pressure (BP) monitoring is essential for timely therapeutic intervention, particularly in patients undergoing major surgery. Among invasive BP measurement sites, the radial artery is commonly used due to its accessibility and ease of catheterization. However, physiologically, the radial artery may underestimate central arterial pressure compared to the femoral artery, especially in patients receiving vasopressors or in critical conditions. This discrepancy can lead to overtreatment with vasopressors and associated complications. Current literature on the accuracy of radial versus femoral BP monitoring is outdated and based solely on observational studies. There is a lack of high-quality randomized data to inform clinical guidelines.

Hypothesis: Femoral arterial pressure monitoring, by offering more accurate hemodynamic data, reduces the need for vasopressor support, particularly norepinephrine, compared to radial artery monitoring.

Primary Objective: To compare the effect of femoral versus radial invasive BP monitoring on the proportion of patients requiring norepinephrine from anesthetic induction to postoperative day 7 (D7) following elective cardiac surgery. Norepinephrine treatment is defined by continuous intravenous administration of norepinephrine for more than 1 minute.

Secondary Objectives :

To compare the following outcomes between the two strategies within the first 7 postoperative days: incidence of acute kidney injury (AKI) according to KDIGO criteria, incidence of cardiac complications (arrhythmias requiring treatment, myocardial injury (troponin >99th percentile or >20% rise from baseline), myocardial infarction, cardiogenic shock, cardiac arrest), vaso-inotropic score (VIS), duration of any vasopressor therapy (days), ICU and hospital length of stay (days), all-cause mortality at day 7 and day 30, total duration (hours/days) and maximal dose of norepineprhine therapy, intraoperative hypotension episodes (MAP<65 mmHg > 5 min), incidence of arterial catheter-related complications (hematoma, bleeding, infection, thrombosis, arterial occlusion, malfunction, dislodgement).

Primary Endpoint: The proportion of patients receiving continuous intravenous norepinephrine from anesthesia induction to postoperative day 7.

Secondary Endpoints:

AKI occurrence or need for renal replacement therapy; cardiac complications: atrial/ventricular arrhythmias requirinf treatment, myocardial injury (troponin >99th percentile or >20% rise from baseline), myocardial infarction (biomarker elevation + ECG or echocardiographic abnormalities), cardiogenic shock, cardiac arrest; maximum VIS in the OR, ICU admission, and day 1; intraoperative hypotension episodes (MAP<65 mmHg > 5 min); total norepinephrine support duration (in hours); duration of any vasopressor therapy; arterial line complications: malfunction, dislodgement, hematoma, thrombosis, infection, bleeding, arterial occlusion; ICU and hospital length of stay (days); all-cause mortality at day 7 and day 30

Study Design: A prospective, multicenter (Besançon and Dijon University Hospitals), randomized, superiority, single-blind, intention-to-treat clinical trial in adults undergoing elective cardiac surgery. Patients are randomized to femoral or radial artery catheterization for continuous BP monitoring.

Sample Size: Based on an expected norepinephrine use rate of 70%, a 15% absolute risk reduction, α = 0.05, and power = 90%, 162 patients per group are required. Accounting for 5% data loss, 340 patients will be enrolled.

Study Arms:

Radial group: invasive BP monitoring via radial artery catheterization Femoral group: invasive BP monitoring via femoral artery catheterization The arterial line is placed under ultrasound guidance in the operating room and maintained postoperatively in the ICU or critical care unit until no longer clinically indicated.

Eligibility Criteria Inclusion: adults patients ≥18 years undergoing elective on-pump cardiac surgery with informed consent.

Exclusion: emergency surgery, use of dual arterial lines, heart transplantation, mechanical circulatory support, contraindications to radial/femoral catheterization, legal or ethical inability to consent.

Study Timeline Inclusion period: 36 months Patient follow-up: 7 days post-surgery Total study duration: 36 months

Data Collection: Clinical data are collected by research staff using an electronic case report form (e-CRF) via CleanWeb™ software.

Expected Impact: There are currently no guidelines specifying the optimal site for invasive BP monitoring. This study aims to provide robust evidence on whether femoral BP monitoring improves clinical outcomes, reduces vasopressor use, and minimizes adverse events. Positive findings could inform future practice guidelines and lead to broader investigations in other clinical settings.

DETAILED DESCRIPTION:
Acute circulatory failure or shock-typically characterized by arterial hypotension-is a major cause of ICU admission and a significant contributor to postoperative complications in surgery. This condition may result from various pathophysiological mechanisms such as arterial vasodilation, hypovolemia, or low cardiac output, frequently triggered by sepsis, inflammation, surgery, or hemorrhage. Hypotension leads to hypoperfusion of vital organs (kidney, brain, heart), significantly increasing patient morbidity and mortality. Consequently, numerous studies have focused on identifying critical blood pressure thresholds and optimizing therapeutic strategies to reduce associated organ dysfunction and mortality.

A key challenge in the management of hypotension is the accuracy of blood pressure (BP) measurement. In clinical practice, invasive arterial pressure is commonly monitored at radial, brachial, or femoral sites. The radial artery is often preferred for its accessibility and ease of catheterization. However, from a physiological standpoint, the radial artery's small diameter and peripheral location can result in discrepancies when compared to central aortic pressure-the actual pressure driving organ perfusion.

Several studies have shown that in states of shock or acute circulatory failure, radial artery pressure measurements often underestimate actual blood pressure compared to more central measurements such as femoral artery pressure. This difference is particularly pronounced in specific physiological and pathological conditions-e.g., during vasoconstrictor use-where systolic pressure gradients between radial and femoral sites may be significant.

As such, accurate blood pressure monitoring is critical in anesthesia and critical care to guide fluid resuscitation, vasopressor therapy, and interpretation of hemodynamic monitoring tools. Inaccurate measurements may lead to excessive exposure to hypotension or unnecessary administration of vasopressors, both of which carry associated risks.

Scientific literature comparing radial and femoral arterial BP monitoring is limited, outdated (mainly from the 1990s), and largely based on observational data. It is well-established that radial artery monitoring can lead to spuriously low BP readings, resulting in inappropriate hemodynamic management, including excessive fluid resuscitation or vasopressor administration.

Observational studies consistently report the following findings:

A systematic pressure gradient (at least 5-10 mmHg in mean arterial pressure) between femoral and radial sites.

The radial site underestimates femoral BP, and thus organ perfusion pressure. This gradient is more pronounced in critically ill patients, particularly those receiving vasopressors, women, or those with severe illness (e.g., refractory shock, sepsis).

These discrepancies in BP measurement are associated with overuse of hemodynamic drugs. Previous studies reported that over one-third of patients had a significant BP gradient between radial and femoral sites-often leading to excessive vasopressor administration. Other works further support this, indicating higher rates of adverse events, including acute kidney injury (AKI), and excessive vasopressor use in patients monitored at the radial site versus the femoral site.

AKI, frequently observed during shock or in surgical patients, is a key concern. In its severe form, it increases operative mortality by 3 to 8 times, lengthens ICU and hospital stays, and dramatically increases healthcare costs. Even mild AKI is a major predictor of long-term outcomes, particularly chronic kidney disease. The kidney is especially vulnerable to both hypotension and excessive vasopressor use. Multiple perioperative and ICU studies have demonstrated correlations between norepinephrine exposure (dose and duration) and increased AKI incidence.

Despite the importance of accurate BP measurement, the debate regarding the optimal site for arterial monitoring remains unresolved. Radial catheterization is less invasive and easier to perform but may result in excessive vasopressor use and associated complications. In contrast, femoral arterial monitoring may offer more precise pressure readings and thereby improve the safety and efficiency of hemodynamic optimization in critically ill or surgical patients.

The central hypothesis of this study is that invasive arterial pressure monitoring at the femoral site is associated with a reduced number of patients requiring vasopressor therapy (e.g., norepinephrine), compared to monitoring at the radial site.

While clinical guidelines address central venous access and the use of ultrasound guidance, no current recommendations specify the optimal arterial site for BP monitoring, primarily due to a lack of high-quality evidence. This study aims to fill that gap, focusing on a routine clinical practice-arterial pressure monitoring in perioperative and critical care settings.

A better understanding of the clinical implications of the measurement site could lead to more precise recommendations for invasive BP monitoring and improve patient care. Results from this trial may influence: the choice of arterial catheterization site, the use and duration of vasopressor therapy, the incidence of renal and cardiovascular complications.

Should this study demonstrate that femoral arterial monitoring improves clinical outcomes, it could lead to changes in clinical practice guidelines and initiate larger-scale investigations in various other critical care and surgical populations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years
* Scheduled cardiac surgery with cardiopulmonary bypass (time between anesthesia consultation and surgery > 48 hours)
* ASA physical status ≥II
* Affiliation with or beneficiary of the French national health insurance system
* Signed informed consent indicating that the participant has understood the purpose and procedures of the study and agrees to participate and comply with its requirements and restrictions

Exclusion Criteria:

* Emergency surgery (before the next working day after decision to operate)
* Surgery requiring the use of two arterial pressure monitoring sites: e.g., aortic arch surgery, aortic dissection, etc.
* Heart transplantation surgery
* Mechanical circulatory support
* Contraindication to radial artery catheterization: failed Allen test, Raynaud syndrome, Buerger disease, major hyperlipidemia
* Contraindication to femoral artery catheterization: puncture of vascular prosthetic material in the femoral area (e.g., femoral bypass, femoral stenting, femoral trifurcation endarterectomy, femoral angioplasty)
* Pregnant or breastfeeding women
* Persons deprived of liberty by judicial or administrative decision; persons under compulsory psychiatric care; persons admitted to a healthcare or social institution for reasons other than research
* Adults under legal protection measures (guardianship, trusteeship, or legal safeguard) or unable to give informed consent
* Subjects currently under exclusion period of another clinical trial or listed in the national registry of research volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with continuous intravenous norepinephrine | Within 7 days after surgery
  Number of patients treated with continuous intravenous norepinephrine to treat arterial hypotension related to vasoplegic syndrome from the time of anesthetic induction until postoperative day 7.
  Norepinephrine treatment is defined by continuous intravenous administration of norepinephrine for more than 1 minute.

SECONDARY OUTCOMES:
Rate of renal complications | Within 7 days after surgery
  Rate of renal complications defined as acute kidney injury according to the KDIGO criteria and/or the need for renal replacement therapy
Rate of cardiac complications | Within 7 days after surgery
  Rate of cardiac complications including: arrhythmias requiring treatment (atrial fibrillation, atrial flutter, ventricular tachycardia, ventricular fibrillation), myocardial injury (defined by an elevation of troponin I or T >99 percentile of the upper reference limit or >20% from the preoperative value), myocardial infarction (defined by elevated cardiac enzymes [cardiac troponin or high-sensitivity cardiac troponin] associated with new Q waves and/or wall motion abnormalities on echocardiography), cardiogenic shock (requiring inotropic support), cardiac arrest
Maximum vasoactive-inotropic score (VIS) | Intraoperatively, during the surgery, from surgical incision to end of surgery, in the operating room
  Higher value of the vasoactive-inotropic score (VIS) (VIS = Dopamine (μg/kg/min) + Dobutamine (μg/kg/min) + 100 × Epinephrine (μg/kg/min) + 100 × Norepinephrine (μg/kg/min) + 10 × Milrinone (μg/kg/min) + 10,000 × Vasopressin (U/kg/min) + 100 × Phenylephrine (μg/kg/min)
Vasoactive-inotropic score (VIS) value | At admission in the postoperative intensive care unit (ICU) (up to 2 hours after surgery)
  Value of the vasoactive-inotropic score (VIS) (VIS = Dopamine (μg/kg/min) + Dobutamine (μg/kg/min) + 100 × Epinephrine (μg/kg/min) + 100 × Norepinephrine (μg/kg/min) + 10 × Milrinone (μg/kg/min) + 10,000 × Vasopressin (U/kg/min) + 100 × Phenylephrine (μg/kg/min)
Maximum vasoactive-inotropic score (VIS) value | Within 1 day after surgery
  Higher value of the vasoactive-inotropic score (VIS) (VIS = Dopamine (μg/kg/min) + Dobutamine (μg/kg/min) + 100 × Epinephrine (μg/kg/min) + 100 × Norepinephrine (μg/kg/min) + 10 × Milrinone (μg/kg/min) + 10,000 × Vasopressin (U/kg/min) + 100 × Phenylephrine (μg/kg/min)
Maximal dose of norepinephrine therapy | Within 7 days after surgery
  Higher rate of norepinephrine infused, expressed in µg/kg/min
Rate of intraoperative hypotension episodes | Intraoperatively, during the surgery, from surgical incision to end of surgery, in the operating room
  Rate of intraoperative hypotensive episodes, defined as a mean arterial pressure (MAP) < 65 mmHg for at least 5 minutes
Cumulative duration of norepinephrine support | Within 7 days after surgery
  Total cumulative duration of norepinephrine support, expressed in hours.
Cumulative duration of any vasopressor therapy | Within 7 days after surgery
  Total cumulative duration of any vasopressor therapy, expressed in hours
Rate of complications related to arterial catheterization and invasive arterial pressure monitoring | Within 7 days after surgery
  Complications related to invasive arterial pressure monitoring including: catheter placement failure, device malfunction, hematoma or bleeding at the insertion site, arterial thrombosis and/or occlusion, and arterial site infection
ICU length of stay | Within 30 days after surgery
  Total cumulative duration of ICU stay from the date of surgery (Day 0) up to postoperative Day 30, inclusive.
Hospital length of stay | Within 30 days after surgery
  Total cumulative duration of hospital stay from the date of surgery (Day 0) up to postoperative Day 30, inclusive.
Mortality | Within 7 and 30 days after surgery
  Day 7 and Day 30 mortality

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Besch, M.D., Ph.D., Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Dijon, Dijon

IPD SHARING:
Plan to Share IPD: No
The protocol will be published. The French legislation did not allow for IPD.

REFERENCES:
- [Derived] Guinot PG, Bronnert R, Grelet T, Bouhemad B, Nguyen M, Besch G; FERARI study group. Femoral versus radial arterial pressure monitoring in cardiac surgery patients: protocol for a randomised controlled multicentric superiority trial (FERARI). BMJ Open. 2026 Jan 28;16(1):e111663. doi: 10.1136/bmjopen-2025-111663. PMID 41605595